CLINICAL TRIAL: NCT02799940
Title: Abnormalities in Lung Computed Tomography and Physiological Alterations in Patients With Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Hospital Regional Rio Gallegos (Other)
Responsible Party: Sponsor
Other Study IDs: MJL001
Record Dates: First submitted 2016-06-02; First posted 2016-06-15 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Computed tomography in acute respiratory distress syndrome: The lung on computed tomography (CT) in patients with acute respiratory distress syndrome (ARDS) has revealed a heterogeneous pattern of lung injury, with areas of normal lung interspersed with altered regions: ground-glass opacification and consolidation among the most frequent. It has been performed quantitative assessments of ARDS by means of CT, thus enabling a correlation of such pathologic details with physiologic, clinical parameters and with patient outcomes. Therefore, the primary objective of the study is to determine the correlation between the extent of oxygenation (PaO2/FiO2) and the degree of consolidation (total CO) in the CT. The secondary objectives are to determine: the correlation between the driving pressure, ventilator variables and the total CO; the independent variables associated with total CO; differences in the CT with respect to the total lung-disease score (total CO plus total value of ground-glass opacification) between survivors and nonsurvivors.

SUMMARY:
The objective of the study is to determine the correlation between the physiological variables and the degree of consolidation in lung computed tomography in patients with acute respiratory distress syndrome

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) involves respiratory failure from different causes, but with a common pathologic manifestation in the form of inflammatory pulmonary edema. Histopathological examination of tissue obtained from patients with ARDS suggests that the pathology is heterogeneous and involves 3 phases: exudative, inflammatory, and fibroproliferative. Such alterations are associated with a decreased lung compliance leading to an increased pressure in the airways under mechanical ventilation (MV) that becomes more pronounced with increasing severity of ARDS, so that the consequent respiratory mechanics has thus been shown to be determinant of patient outcomes. In addition, computed tomography (CT) has revealed a heterogeneous pattern of lung injury, with areas of normal lung interspersed with morphologically altered regions, among which abnormalities the ground-glass opacification and consolidation are the most frequent. It has been performed quantitative assessments of ARDS by means of CT, thus enabling a correlation of such pathologic details with physiologic and clinical parameters as well as with patient outcomes. From the above, the investigators hypothesize that in patients with ARDS, a greater involvement in oxygenation and higher mechanical alterations will be correlated with a more advanced consolidation in the CT scan. Therefore, the primary objective of the study will be to determine the correlation between the extent of oxygenation (assessed by the PaO2/FiO2 ratio) and the degree of consolidation (total CO) in the CT scan. The secondary objectives will be: (1) to determine the correlation between the driving pressure and the total CO as evidenced by CT; (2) to determine the correlation between the static pressure and the total CO; (3) to determine the correlation between the static compliance and the total CO; (4) to determine the correlation between oxygenation index and the total CO; (5) to determine the correlation between the lung injury score (LIS) and the total CO; (6) to determine the correlation between ventilator free days and the total CO; (7) to determine the independent variables associated with total CO; (8) to determine differences in the CT with respect to the total lung-disease score [total CO plus total value of ground-glass opacification (total GC)] between survivors and nonsurvivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients 15 years of age or older who have been receiving MV and have been defined as with ARDS according to the Berlin definition

Exclusion Criteria:

Patients with chronic pulmonary disease, with an expected duration of MV shorter than 48 h, or with a high risk of death within 3 months for reasons other than ARDS as well as patients having made the decision to withhold life-sustaining treatment along with those exhibiting clinical instability that could not be moved to the radiology department in order to perform CT scans.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 15 years of age or older admitted in the intensive care unit (ICU) of the Rio Gallegos Regional Hospital who have been receiving MV and have been defined as with ARDS according to the Berlin definition.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-08; Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

PRIMARY OUTCOMES:
Correlation between the extent of oxygenation and the degree of consolidation (total CO) in the CT scan. | Within the first 60 days (plus or minus 3 days) after admission to Hospital
  The extent of oxygenation will be assessed by the PaO2/FiO2 ratio obtained the day of diagnosis of ARDS

SECONDARY OUTCOMES:
Correlation between the driving pressure and the total CO as evidenced by CT | Within the first 60 days (plus or minus 3 days) after admission to Hospital
  The driving pressure will be obtained over the first 24 hours after randomization
Correlation between the static pressure and the total CO evidenced by CT | Within the first 60 days (plus or minus 3 days) after admission to Hospital
  The static pressure will be obtained over the first 24 hours after randomization
Correlation between the static compliance and the total CO evidenced by CT | Within the first 60 days (plus or minus 3 days) after admission to Hospital
  The static compliance will be obtained over the first 24 hours after randomization
Correlation between oxygenation index and the total CO evidenced by CT | Within the first 60 days (plus or minus 3 days) after admission to Hospital
  The oxygenation index will be obtained over the first 24 hours after randomization
Correlation between the lung injury score (LIS) and the total CO evidenced by CT | Within the first 60 days (plus or minus 3 days) after admission to Hospital
  The lung injury score (LIS) will be obtained over the first 24 hours after randomization
Correlation between ventilator free days and the total CO evidenced by CT | Within the first 60 days (plus or minus 3 days) after admission to Hospital
Independent variables associated with total CO | Within the first 60 days (plus or minus 3 days) after admission to Hospital
  A multivariate logistic-regression model will be used to independent assess variables that showed correlation with total CO. The investigators also will be introduced in the model the potential confounders: age, gender, APACHE-II score and SOFA score.
Differences in the CT with respect to the total lung-disease score [total CO plus total value of ground-glass opacification (total GC)] between survivors and nonsurvivors. | Within the first 60 days (plus or minus 3 days) after admission to Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Santa Cruz, Doctor, Principal Investigator — Hospital Regional Rio Gallegos
Locations (1):
- Hospital Regional Rio Gallegos, Río Gallegos, Santa Cruz Province, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoenfeld DA, Bernard GR; ARDS Network. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of treatments for acute respiratory distress syndrome. Crit Care Med. 2002 Aug;30(8):1772-7. doi: 10.1097/00003246-200208000-00016. PMID 12163791
- [Result] Ware LB, Matthay MA. The acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1334-49. doi: 10.1056/NEJM200005043421806. No abstract available. PMID 10793167
- [Result] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Result] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Result] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Result] Maunder RJ, Shuman WP, McHugh JW, Marglin SI, Butler J. Preservation of normal lung regions in the adult respiratory distress syndrome. Analysis by computed tomography. JAMA. 1986 May 9;255(18):2463-5. PMID 3701964
- [Result] Desai SR, Wells AU, Rubens MB, Evans TW, Hansell DM. Acute respiratory distress syndrome: CT abnormalities at long-term follow-up. Radiology. 1999 Jan;210(1):29-35. doi: 10.1148/radiology.210.1.r99ja2629. PMID 9885583
- [Result] Gattinoni L, Pesenti A, Bombino M, Baglioni S, Rivolta M, Rossi F, Rossi G, Fumagalli R, Marcolin R, Mascheroni D, et al. Relationships between lung computed tomographic density, gas exchange, and PEEP in acute respiratory failure. Anesthesiology. 1988 Dec;69(6):824-32. doi: 10.1097/00000542-198812000-00005. PMID 3057937
- [Result] Burnham EL, Hyzy RC, Paine R 3rd, Kelly AM, Quint LE, Lynch D, Curran-Everett D, Moss M, Standiford TJ. Detection of fibroproliferation by chest high-resolution CT scan in resolving ARDS. Chest. 2014 Nov;146(5):1196-1204. doi: 10.1378/chest.13-2708. PMID 24722949
- [Result] Owens CM, Evans TW, Keogh BF, Hansell DM. Computed tomography in established adult respiratory distress syndrome. Correlation with lung injury score. Chest. 1994 Dec;106(6):1815-21. doi: 10.1378/chest.106.6.1815. PMID 7988207
- [Result] Murray JF, Matthay MA, Luce JM, Flick MR. An expanded definition of the adult respiratory distress syndrome. Am Rev Respir Dis. 1988 Sep;138(3):720-3. doi: 10.1164/ajrccm/138.3.720. No abstract available. PMID 3202424
- [Result] Goodman LR, Fumagalli R, Tagliabue P, Tagliabue M, Ferrario M, Gattinoni L, Pesenti A. Adult respiratory distress syndrome due to pulmonary and extrapulmonary causes: CT, clinical, and functional correlations. Radiology. 1999 Nov;213(2):545-52. doi: 10.1148/radiology.213.2.r99nv42545. PMID 10551239
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Result] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069